CLINICAL TRIAL: NCT04339855
Title: Artificial Intelligence Combined With LCI for Colorectal Polyp Detection
Brief Title: AI for Colorectal Polyp Detection in Endoscopy
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Johannes Gutenberg University Mainz (Other)
Responsible Party: Principal Investigator, Prof. Helmut Neumann, Director Interdisciplinary Endoscopy, Johannes Gutenberg University Mainz
Other Study IDs: HN_01KR7Zt
Record Dates: First submitted 2020-04-07; First posted 2020-04-09 (Actual); Last update posted 2020-09-07 (Actual); Status verified 2020-09

CONDITIONS: Focus of the Study is to Evaluate a New Developed Deep-learning Computer-aided Detection System in Combination With LCI for Colorectal Polyp Detection

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: CAD with LCI for colorectal polyp detection — Polyps within fully recorded endoscopy videos with LCI mode, covering the whole spectrum of adenomatous histology, are used to evaluate the efficacy of CAD with LCI for polyp detection.

SUMMARY:
Linked color imaging (LCI) has shown its effectiveness in multiple randomized controlled trials for enhanced colorectal polyp detection. Most recently, artificial intelligence (AI) with deep learning through convolutional neural networks has dramatically improved and is increasingly recognized as a promising new technique enhancing colorectal polyp detection. Study aim was to evaluate a new developed deep-learning computer-aided detection (CAD) system in combination with LCI for colorectal polyp detection.

ELIGIBILITY:
Inclusion Criteria:

* Full endoscopy withdrawal videos with LCI of patients ondergoing screening or surveillance endoscopy

Exclusion Criteria:

* non adequate bowel preparation
* no full length withdrawal in LCI mode

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients ondergoing screeining or surveillance endoscopy
Sampling Method: Non-Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2019-02-01 (Actual); Primary Completion 2020-08-31 (Estimated); Study Completion 2020-09-30 (Estimated)

PRIMARY OUTCOMES:
Colorectal polyp detection rate in comparison to traditional detection rate | 2019-2020

CONTACTS AND LOCATIONS:
Overall Officials: Helmut Neumann, Prof. Dr., Principal Investigator — Head of Interdisciplinary Endoscopy
Locations (1):
- University Hospital Mainz, Mainz, Germany

IPD SHARING:
Plan to Share IPD: Undecided